CLINICAL TRIAL: NCT05544214
Title: An Open Label, Randomized, Single Dose Crossover Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD 371 in Healthy Subjects
Brief Title: Clinical Study to Evaluate the Pharmacokinetics, Safety and Tolerability of CKD 371 in Healthy Subjects
Acronym: CKD-371
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A127_01BE2206
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-09

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): Period 1 - A single dose of 2 tablets(D745, D759) under fasting condition.
  Period 2 - A single dose of 1 tablets(CKD-371) under fasting condition.
  Interventions: Drug: CKD-371
- Sequence 2 (Experimental): Period 1 - A single dose of 1 tablets(CKD-371) under fasting condition.
  Period 2 - A single dose of 2 tablets(D745, D759) under fasting condition.
  Interventions: Drug: CKD-371

INTERVENTIONS:
Drug: CKD-371 — PO
  Other Names: D745, D759

SUMMARY:
This study is an open-label, randomized, single dose, crossover study to evaluate the pharmacokinetics, safety and tolerability of CKD-388 in healthy subjects

DETAILED DESCRIPTION:
To healthy 32 subjects, following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

Reference drug: D745, D759 / Test drug: CKD-371

Pharmacokinetic blood samples are collected up to 48hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults volunteers aged between 19 and 45 years old at the time of screening
2. Weight ≥50kg, with calculated body mass index (BMI) of 18.0 to 29.9 kg/m2 at the time of screening
3. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial

Exclusion Criteria:

1. Those with clinically significant diseases or history in cardiovascular system, respiratory system, liver, kidney, hematological, gastrointestinal, endocrine system, immune system, skin system, mental/nervous system, etc
2. Those who have symptoms of acute disease within 28 days of the the first dose of the investigational product
3. Those who with a history of influencing drug absorption, distribution, metabolism, and excretion
4. Those who have a hypersensitivity reaction or a history of clinically significant hypersensitivity reaction or a history of drug abuse inculding SGLT2 inhibitor class component or DPP 4 inhibitor class or same class component drugs containing ingredients
5. Those with clinically significant active chronic disease
6. Those with genetic problems such as galactose intolerance, Lapp lactase deficiency or glucose galactose malabsorption
7. A person who has had one or more of the following results in screening tests including re-examination

   * AST, ALT > UNL (upper normal limit) x 2.5
   * Fasting glucose < 70 mg/dL
   * Calculated by Cockcroft Gault formula Creatinine clearance is 75mL/min or less (Cockcroft Gault GFR = (140 age) * (Wt in kg) / (72 * Cr))
   * QTc > 470 msec as a result of ECG
   * Urine-hCG test is positive(if it is limited to female subjects)
8. Those who test positive for HBs Ag, HCV Ab, HIV Ab, or VDRL
9. Those who have taken prescription medicine (ETCs), including prescription drugs, within 14 days of the first dose
10. Those who have taken over-the-counter medicines (OTC) including herbal medicines within 7 days of the first dose
11. Clinically significant allergic diseases, mild allergic rhinitis that do not require medication, and allergic dermatitis can be selected
12. Those who cannot eat the standard meal provided by the institution
13. Those who donated whole blood within 60 days prior to the first dose or donated component blood within 20 days
14. Those who received a blood transfusion within 30 days prior to the first dose
15. Those who have participated in other clinical studies or bioequivalence studies within 6 months of the first dose and administered the investigational drug
16. Those who had taken any drug known as a strong inducer or inhibitor of drug-metabolizing enzymes within 30 days prior to the first dose of the investigational product
17. Those who have continuously consumed grapefruit juice or caffeine > 5 cups a day, or cannot refrain from intake during hospitalization
18. Consistently drinking alcohol > 30 days or unable to abstain from alcohol during hospitalization
19. Excessive smokers > 20 cigarettes non-daily or unable to quit smoking during hospitalization
20. Pregnant or childbearing potential and lactating women
21. Those who consent to the use of reliable contraception(contraceptive methods other than hormones: use of condoms, intrauterine devices (IUD, IUS), tubal ligation, cervical cap, contraceptive diaphragm, etc.) during the clinical trial and not to donate sperm until 2 month after the last administration of investigational product
22. Clinical laboratory test results and other reasons eg, a person who does not respond to requests and instructions, or who judges the investigator to be inappropriate to participate in the clinical trial with a non-cooperative attitude

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-371, D745+D759 | Pre-dose(0hr), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48hr
  Area under the CKD-371, D745+D759 concentration in blood-time curve from zero to final
Cmax of CKD-371, D745+D759 | Pre-dose(0hr), post-dose 0.33, 0.67, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48hr
  The maximum CKD-388/D418 concentration in blood sampling time

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea